CLINICAL TRIAL: NCT07196059
Title: Assessment of Delphinol® Dose on Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Anklam-Extrakt GmbH (Unknown)
Responsible Party: Principal Investigator, Richard Bloomer, Dean of School of Health Studies, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PRO-FY2020-66
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Delphinol; antioxidant; vascular function
MeSH Terms: interventions — Delphinol

STUDY DESIGN:
Intervention Model Description: Participants will receive each of 4 interventions over approximately 8 weeks. On the first day baseline measures will be obtained, and participants will begin the first treatment. For each arm, participants will take the treatment daily for 8 days. They will then return to the lab on the 8th day. Participants will then have a "wash out" period of 7 days prior to the start of the next arm.
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 60mg Delphinol® (Experimental): Capsule to be taken daily for 8 days
  Interventions: Dietary Supplement: Delphinol
- 120 mg Delphinol (Experimental): Capsule to be taken daily for 8 days
  Interventions: Dietary Supplement: Delphinol
- 180 mg Delphinol (Experimental): Capsule to be taken daily for 8 days
  Interventions: Dietary Supplement: Delphinol
- Placebo (Placebo Comparator): Capsule to be taken daily for 8 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Delphinol — Contains maqui berry powder
  Arms: 120 mg Delphinol; 180 mg Delphinol; 60mg Delphinol®
Dietary Supplement: Placebo — Contains cellulose
  Arms: Placebo

SUMMARY:
Maqui berry standardized extract (e.g. Delphinol®) has been used with success to modulate blood glucose and associated variables at a dosage of 450mg daily. Lower dosages have also been used with favorable effects. However, it is unknown what dosage is optimal for positively impacting vascular function. The purpose of this study is to determine the impact of Maqui berry standardized extract (e.g. Delphinol®) at varying dosages on vascular function assessed using the perfusion index, Vendys, and blood nitrate/nitrite concentrations.

DETAILED DESCRIPTION:
Antioxidant compounds have been well-studied in relation to surrogate measures of overall health, with a particular impact on the function of blood vessels. Delphinol® is a botanical agent (an extract of maqui berries) with antioxidant properties primarily owing to its high anthocyanin content. Delphinol® has excellent bioavailability, as demonstrated recently. Acute and chronic anthocyanin consumption has demonstrated the ability to improve vascular reactivity assessed via flow-mediated dilation and pulse wave velocity across a range of dosages . Antioxidant compounds have also been reported to favorably impact nitric oxide, often estimated using the surrogate measure of blood nitrate/nitrite.

In a previous study using Delphinol® at various dosages, Delphinol® significantly and dose-dependently improved glucose homeostasis acutely, with noted lowering of blood glucose and lipids. The mechanism of action for this effect appears related to a novel sodium glucose cotransporter inhibition . This favorable effect on glucose and lipid metabolism is an effect that some have suggested may be associated with the protection of vascular function. A dosage of 450mg of Delphinol® daily has resulted in improvements in oxidative stress markers, another factor that can potentially contribute to vascular homeostasis. Together, these studies suggest Delphinol® may influence vascular function; however, no studies have directly determined this in human subjects.

Though similar studies exist demonstrating anthocyanin consumption resulting in improvements in vascular function, none to date have investigated different doses of a maqui extract on vascular function as assessed using the digital thermal monitoring of reperfusion. Digital thermal monitoring is suggested to be a more reliable measure of vascular function because it removes the sonographer variability; that is, accurately capturing the brachial artery with an ultrasound transducer can be very challenging.

The aim of the present study is to determine the impact of Delphinol® at varying dosages on vascular function assessed using the perfusion index, Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring), and blood nitrate/nitrite concentrations in men and women. While it may be logical to assume that the higher dosage may provide a more robust overall effect with regards to our outcome measures, we will maintain a conservative non-directional hypothesis related to dose. That said, we do hypothesize that all doses of the ingredient will result in small improvements in the measured vascular indices.

ELIGIBILITY:
* age 18-35 years
* male or female
* body mass index (BMI) between 18-29.9 kg/m2 (not obese)
* non-smoker
* no diagnosed history of diabetes
* no diagnosed history of cardiovascular disease including any vascular disease
* no diagnosed history of neurological disease
* no consumption of alcohol or fruit within 48 hours of testing
* no consumption of caffeine-containing beverages within at least 48 hours of testing
* 12-lead ECG without significant heart rate and rhythm abnormalities and blood glucose within normal limits (as reviewed by Tara Hunter, BSN and confirmed by Dr. John Hyden, MD as needed)
* if female, not be pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Baseline Perfusion Index | On day 1
  Perfusion index will be measured using a fingertip pulse oximeter prior to first arm of study.
Perfusion Index after 60 mg Delphinol treatment | 90 min post supplement ingestion on day 8 of treatment
  Perfusion index will be measured using a fingertip pulse oximeter on the 8th day of 60 mg Delphinol treatment.
Perfusion Index after 120 mg Delphinol treatment | 90 min post supplement ingestion on day 8 of treatment
  Perfusion index will be measured using a fingertip pulse oximeter on the 8th day of 120 mg Delphinol treatment.
Perfusion Index after 180 mg Delphinol treatment | 90 min post supplement ingestion on day 8 of treatment
  Perfusion index will be measured using a fingertip pulse oximeter on the 8th day of 180 mg Delphinol treatment.
Perfusion Index after placebo treatment | 90 min post supplement ingestion on day 8 of treatment
  Perfusion index will be measured using a fingertip pulse oximeter on the 8th day of placebo treatment.
baseline Vendys II endothelial measure | On day 1
  Endothelial measure will be determined using Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring) prior to first arm of study
Vendys II endothelial measure after 60 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Endothelial measure will be determined using Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring) 90 min post 60 mg Delphinol treatment ingestion
Vendys II endothelial measure after 120 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Endothelial measure will be determined using Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring) 90 min post 120 mg Delphinol treatment ingestion
Vendys II endothelial measure after 180 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Endothelial measure will be determined using Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring) 90 min post 180 mg Delphinol treatment ingestion
Vendys II endothelial measure after placebo treatment | 90 min post supplement ingestion on day 8 of treatment
  Endothelial measure will be determined using Vendys II (a tool to measure endothelial vascular function via digital thermal monitoring) 90 min post placebo treatment ingestion
Baseline Blood nitrate/nitrite | On day 1
  Baseline blood nitrate/nitrite will be determined prior to first arm of study
Blood nitrate/nitrite after 60 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Blood nitrate/nitrite will be determined on 8th day of treatment, 90 min post 60 mg Delphinol treatment ingestion
Blood nitrate/nitrite after 120 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Blood nitrate/nitrite will be determined on 8th day of treatment, 90 min post 120 mg Delphinol treatment ingestion
Blood nitrate/nitrite after 180 mg Delphinol treatment | 90 min post treatment ingestion on day 8 of treatment
  Blood nitrate/nitrite will be determined on 8th day of treatment, 90 min post 180 mg Delphinol treatment ingestion
Blood nitrate/nitrite after placebo treatment | 90 min post treatment ingestion on day 8 of treatment
  Blood nitrate/nitrite will be determined on 8th day of treatment, 90 min post placebo treatment ingestion

SECONDARY OUTCOMES:
Blood pressure | At baseline and on day 8 of each treatment, prior to treatment ingestion
  Resting blood pressure will be measured
Heart rate | At baseline and on day 8 of each treatment, prior to treatment ingestion
  Resting heart rate will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bloomer, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Research, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided